CLINICAL TRIAL: NCT04956848
Title: A Comparison of Two Models Used for Identifying Embryos With the Best Chance of Inducing Pregnancy: A Pilot Study
Brief Title: Comparing KIDScore™ D5 and iDAScore®. The KiDA Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitrolife (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1571 - KiDA
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: IVF; Infertility
Keywords: Embryos; Embryo scoring; Blastocyst selection; Pregnancy rate; Live birth rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: A pilot study randomizing embryos into two study groups comparing two decision support tools in the ranking of embryos for transfer.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embryo selection supported by KIDScore™ D5 (No Intervention): Each embryo reaching at least developmental stage of 3BB will annotated by an embryologist using the parameters required by the KIDScore™ D5. The embryo with the highest KIDScore™ will be selected proposed for transfer.
- Embryo selection supported by iDAScore® (Experimental): Images of all the embryos reaching at least developmental stage of 3BB will be analyzed by iDAScore®. The embryo with the highest iDAScore® will be proposed selected for transfer.
  Interventions: Device: iDAScore®

INTERVENTIONS:
Device: iDAScore® — Images of all the embryos reaching at least developmental stage of 3BB will be analyzed by iDAScore®. The embryo with the highest iDAScore® will be proposed for transfer.
  Arms: Embryo selection supported by iDAScore®

SUMMARY:
A pilot study to gather information on clinical pregnancy rates for preparation of the planning of a larger randomized controlled trial comparing two decision support tools: the deep learning tool iDAScore® and the current annotation model, KIDScore™ D5.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing IVF/ICSI-treatment with controlled ovarian stimulation with gonadotrophins and the intention to treat by transfer of a single day 5 fresh blastocyst on day 5.
2. At least two good quality blastocysts (GQB) on day 5 (3BB or better on the Gardner scale), originating from normally fertilized oocytes (2PN).

Exclusion Criteria:

1. Previous participation in this RCT
2. Concurrent participation in another investigation
3. Intention to perform any form of preimplantation genetic testing
4. Fertility preservation
5. Planned transfer on day 2-4
6. Female age >42 years
7. A reduced likelihood of obtaining two good quality blastocysts on day 5 as evidenced by an AFC <5 (if available, AFC=antral follicle count)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | After 6 weeks of gestation
  Ultrasound evidence of an intrauterine pregnancy with a fetal heart observed

SECONDARY OUTCOMES:
Positive hCG rate per randomized patient | From day 13 following embryo transfer
  An hCG measurement using urinary sticks with a sensitivity of 25 IU/L
Rate of non-viable intrauterine pregnancies per randomized patient | After 6 weeks of gestation
  Ultrasound evidence of an intrauterine pregnancy but with no fetal heart observed
Clinical pregnancy rate in patients with maternal age above 35 | After 6 weeks of gestation
  Ultrasound evidence of an intrauterine pregnancy with a fetal heart observed

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Schmidt, MD, Principal Investigator — Göteborgs IVF klinik
Locations (2):
- Sweden (2):
  - Göteborgs IVF klinik, Gothenburg
  - Fertilitetsenheten, Universitetssjukhuset Örebro, Örebro

IPD SHARING:
Plan to Share IPD: No